CLINICAL TRIAL: NCT05958420
Title: Evaluation of HDL Subfraction Changes and HDL-Associated Enzymes in Liver Failure Patients and Healthy Donors
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İlker Onguc Aycan, Prof. Dr. İlker Öngüç Aycan, Akdeniz University
Other Study IDs: KC-HDL
Record Dates: First submitted 2023-07-06; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Liver Failure
Keywords: Liver Failure; HDL Subfractions; ApoA1; CETP; LCAT
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with liver failure
- Group 2: Healthy donors

SUMMARY:
This study aimed to determine high-density lipoprotein (HDL) subfraction profile and HDL-associated enzyme changes in liver failure patients and healthy donors.

DETAILED DESCRIPTION:
Objectives: This study aimed to determine high-density lipoprotein (HDL) subfraction profile and HDL-associated enzyme changes in liver failure patients and healthy donors.

Materials and Methods: Twenty liver failure patients and twenty healthy donors are selected. Blood samples obtained from all patients prior to transplant will analyzed. HDL subfraction analysis will done by continuous disc polyacrylamide gel electrophoresis. Plasma levels of apolipoprotein A-1 (ApoA-I), cholesteryl ester transfer protein (CETP), and lecithin-cholesterol acyltransferase (LCAT) will determined by enzyme-linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Liver failure patients

Exclusion Criteria:

* patients not giving consent
* Participants who had oncological and hematological diseases, coronary failure, kidney failure, malnutrition, diabetes, traumatic brain injury, or cadaveric LT and who were using psychoactive medicines or having a respiratory system or CNS diseases were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who underwent living donor LT procedure between 2018 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
HDL Subfractions | Blood will collected from all patients before surgery
  Evaluation of HDL Subfractions in groups

SECONDARY OUTCOMES:
HDL-associated enzymes | Blood will collected from all patients before surgery
  ApoA1, CETP and LCAT levels in groups

CONTACTS AND LOCATIONS:
Overall Officials: İlker O Aycan, Study Chair — Akdeniz University
Locations (1):
- AkdenizU, Antalya, Turkey (Türkiye)